CLINICAL TRIAL: NCT04593771
Title: Randomized, Blinded, Single-arm Intradermal Injection, Control of Similar Products on the Market, the Safety Pre-evaluation Phase I Clinical Trial of BCG-PPD in Healthy People
Brief Title: Phase I Clinical Protocol of BCG-PPD in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Sichuan Center for Disease Control and Prevention (Other Government); Neijiang Center for Disease Control and Prevention (Unknown); Beijing Kangterike Statistical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: LKM-2020-PPD01
Record Dates: First submitted 2020-09-27; First posted 2020-10-20 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Tuberculosis
Keywords: diagnosis of tuberculosis; epidemiological investigation of tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The statistician and the blind operators who do not participate in the trial will perform drug blinding,stick the printed drug label on the designated position of each drug according to the blind bottom. After completing the blind programming, the blind bottom will be sealed and handed over to the sponsor. The blind editors shall not participate in other related work of this clinical trial, and shall not disclose to any personnel participating in the trial.Subjects were randomly injected intracutaneously with BCG-PPD test drugs or BCG-PPD control drugs.All subjects, some investigators and other staff participating in the study were kept blind.The investigators designated in the study to extract drugs are non-blind personnel, and are not allowed to disclose the subject's grouping and skin test information to others, nor are they allowed to participate in any other procedures in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 80 healthy people were randomly assigned to the experimental group and the control group. The experimental group was injected with BCG-PPD once.
  Interventions: Drug: BCG-PPD
- control group (Other): 80 healthy people were randomly assigned to the experimental group and the control group. The control group was injected with BCG-PPD was marketed once.
  Interventions: Drug: BCG-PPD

INTERVENTIONS:
Drug: BCG-PPD — BCG-PPD was used for skin test in 40 healthy people, and BCG-PPD was marketed in other 40 healthy people (as control)

SUMMARY:
A total of 80 healthy people aged 65 years and below who are randomly assigned to the experimental group and the control group. The experimental group is injected with BCG-PPD test drug once, and the control group is injected with BCG-PPD control drug once.Subjects will undergo physical examination, vital signs, blood routine, urine routine, blood biochemistry, electrocardiogram, HIV antibody test and blood pregnancy test for women of childbearing age during the screening period.Vital signs were checked before skin test, the injection site was photographed at 0min after skin test, and vital signs were checked at 30min after skin test.Vital signs examination, injection site photography and injection site reaction measurement were performed 48h and 72h after skin test.Physical examination, vital signs, routine blood test, routine urine test, biochemical test, electrocardiogram and blood pregnancy test of women of childbearing age were performed again 7 days after skin test to evaluate the safety of BCG-PPD.

DETAILED DESCRIPTION:
Prior to the commencement of the study, the Investigator/his authorized officer will contact the subject and/or guardian to enroll the candidate subjects and invite them to participate in the study.Subjects who are eligible for screening receive the drug number in the order they arrive at the random number allocation room.During the screening period, physical examination, vital signs, blood routine, urine routine, blood biochemistry, electrocardiogram, HIV antibody test and blood pregnancy test (only women of childbearing age).Inverstigator absorb and inject 0.1ml drug into the upper and middle 1/3 of the left forearm by Mondo's method. The reaction of the injection site was checked and photographed at 0min, 48h and 72h after the skin test. Meanwhile, the transverse and longitudinal diameers of skin induration and redness were measured at 48h and 72h after the skin test.Vital signs are checked at 30min after skin test.Vital signs examination, injection site photography and reaction measurement are performed 48h and 72h after skin test.Physical examination, vital signs, routine blood test, routine urine test, biochemical test, electrocardiogram and blood pregnancy test are performed again 7 days after skin test.All AE occurred within 7 days after skin test were recorded by a diary card. AE related to the test drug should be followed up to the end of the event.Skin test of subjects aged 18-45 years shall be conducted first. After safety assessment, skin test of subjects aged 46-65 years old, 6-17 years old and under 6 years old shall be conducted successively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-65 (including 65 years old), male and female.
2. I (and/or my guardian) agree to participate in the study and sign the informed consent.
3. I (and/or guardian) can comply with the requirements of the clinical trial protocol to participate in the follow-up.
4. No history of tuberculosis, family history of tuberculosis, and history of close contact with tuberculosis (refers to direct contact with registered tuberculosis patients from 3 months before their diagnosis to 14 days after the start of anti-tuberculosis treatment).
5. No pulmonary or external tuberculosis, and no respiratory symptoms or other systemic symptoms of tuberculosis.
6. Medical history of careless, liver, kidney, digestive tract, nervous system, mental and metabolic abnormalities after signing the informed consent.
7. Vital signs (body temperature (axillary temperature) < 37.3℃, blood pressure (people aged 18 and over: systolic blood pressure < 140mmHg, diastolic blood pressure < 90mmHg);People aged 6 to 17: systolic blood pressure < 120mmHg, diastolic blood pressure < 80mmHg;No abnormal blood pressure, pulse rate 50 ~ 100 times /min, electrocardiogram, physical examination or abnormality has no clinical significance.
8. Laboratory tests, including blood routine, urine routine and blood biochemical tests, showed no abnormalities or abnormalities had no clinical significance.

Exclusion Criteria:

1. Patients with acute infectious diseases (such as measles, pertussis, influenza, pneumonia, etc.), acute ophthalmic membranitis, acute otitis media, generalized skin diseases and allergic constitution (people with allergy history to two or more drugs or foods, or known allergy and scar constitution to this drug component)
2. Subjects have any serious disease, such as: tumor, progressive atherosclerosis or diabetes with complications, chronic obstructive pulmonary disease requiring oxygen therapy, acute or progressive liver or kidney disease, congestive heart failure, etc.
3. A history of convulsion, epilepsy, mental illness and/or a family history of mental illness.
4. is known or suspected (or has a high risk might) damage or abnormal immune function, such as immune inhibitors or immune enhancer treatment, in 3 months to accept glucocorticoid, outside of the gastrointestinal tract immunoglobulin preparations or blood products or plasma extract, human immunodeficiency virus infection or related diseases.
5. The test results of human immunodeficiency virus (HIV) antibody are positive
6. Before enrollment, the interval between inoculation of live attenuated vaccine is less than 28 days, and the interval between inoculation of other vaccines is less than 14 days
7. In the acute stage of disease or acute onset of chronic disease (3 days before skin test)
8. Is participating in or has participated in any other clinical investigator within 3 months prior to this clinical study
9. pregnant or lactating women, or planning to become pregnant during the study period.
10. On-site inquiry for drug abuse and alcohol abuse.
11. Persons with upper extremity disabilities
12. Birth weight less than 2.5kg, or premature and difficult birth (for infants under one year of age)
13. Newborn with respiratory distress syndrome, pathological jaundice, congenital malformations, developmental disorders and congenital diseases (for infants under 1 year of age)
14. The investigator believes that there are any conditions such as poor compliance that may affect the evaluation of the trial.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Evaluate the incidence of all adverse event and results of laboratory tests | 7 days after injection
  Record and evaluate the incidence of all adverse event within 7 days after injection；Record and evaluate abnormal incidence of blood routine, urine routine, blood biochemical and electrocardiogram indicators 7 days after injection
Evaluate the effectiveness of the product by measuring the size of the skin response | 48 to 72 hours after injection
  The transverse and longitudinal diameters (millimetre) of skin induration and redness, as well as local double circles, blisters, necrosis, and lymphangitis, were recorded at 48h and 72h after injection

CONTACTS AND LOCATIONS:
Overall Officials: Ting Huang, Master, Principal Investigator — Sichuan Center for Disease Control and Prevention
Locations (1):
- Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan, China